CLINICAL TRIAL: NCT00834158
Title: Efficacy of Sequential Arterial and Portal Vein Embolizations on Increasing the Resectability of Hepatitis B Related Primary Hepatocellular Carcinoma
Brief Title: Efficacy of Sequential TACE and PVE on the Resectability of Hepatitis B Related HCC
Acronym: TACEPVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-006
Record Dates: First submitted 2009-01-31; First posted 2009-02-03 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatitis B; Transarterial chemoembolization (TACE); Portal vein embolization (PVE); Surgical resection; Disease-free survival; Overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE (Active Comparator): perform TACE only
  Interventions: Procedure: TACE
- TACE+PVE (Experimental): perform TACE and PVE sequentially
  Interventions: Procedure: TACE; Procedure: PVE

INTERVENTIONS:
Procedure: TACE — 1 time
  Other Names: transaterial chemoemblization
Procedure: PVE — 1 time
  Other Names: portal vein embolization
  Arms: TACE+PVE

SUMMARY:
A primary hepatocellular carcinoma (HCC) is generally regarded as unresectable if the future liver remnant (FLR)≤40％ of total liver volume in patient with underlying liver disease, such as hepatitis B. In China, TACE is the most common treatment for these unresectable HCC. Recently, PVE has been employed to enlarge the FLR of the patients so as to increase the resectability and surgical safety of major hepatectomies. In order to shut the arterio-portal shunt in the liver and control the tumor progress TACE sometimes is performed before PVE. In this study we design a randomized control trial to investigate the efficacy of sequential TACE and PVE on increasing the resectability of hepatitis B related HCC compared with TACE alone.

DETAILED DESCRIPTION:
In China, primary hepatocellular carcinoma (HCC) is mostly a hepatitis B related disease. The liver function of these patients has been damaged, which often limit the execution of major hepatectomy. A tumor is generally regarded as unresectable if the future liver remnant (FLR)≤40％ of total liver volume in patient with underlying liver disease. In China, TACE is the most common treatment for these unresectable HCC. TACE can slow down tumor progress but has little effect on enlarging FLR. Recently, PVE has been employed to enlarge the FLR of the patients so as to increase the resectability and surgical safety of major hepatectomies. But the intrahepatic arterioportal shunt and the tumor progress has decreased the effect of PVE. In order to shut the arterioportal shunt and control the tumor progress TACE sometimes is performed before PVE. In this study we design a randomized control trial to investigate the efficacy of sequential TACE and PVE on increasing the resectability of hepatitis B related HCC compared with TACE alone.

ELIGIBILITY:
Inclusion Criteria:

1. age:20-65years old;
2. with a clinical diagnosis of primary liver cancer, with HBsAg positive,without any therapy for tumor;
3. single lesion with a diameter >6.5cm,or multiple lesions locating within half liver or adjacent three lobe;
4. estimated liver remnant volume ≤40%
5. with a liver function of Child-Pugh class A,and ALT≤80IU/l.

Exclusion criteria:

1. reject to attend；
2. portal vein trunk has been compressed by tumor;
3. diffuse type cancer or with extensive cancer thrombus in main branches of PV,HV,IVC or bile duct;
4. with extrahepatic metastasis;
5. with obvious portal hypertension (with moderate to severe varix in esophagus and/or gastric fundus, enlarged spleen,WBC<4×109／L, PLT<80×109／L)
6. with diabetes
7. allergy to iodine

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
the rate of tumor resection after intervention | 1 to 2 months

SECONDARY OUTCOMES:
rate of survival | 1, 3, 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, China